CLINICAL TRIAL: NCT03873012
Title: Determination of the Duration of the Dual Antiplatelet Therapy by the Degree of the Coverage of The Struts on Optical Coherence Tomography From the Randomized Comparison Between Everolimus-eluting Stents Versus Biolimus A9-eluting Stents: Retrospective and Prospective Follow-up Study for Patients Who Were Enrolled in the Previous DETECT-OCT Study
Brief Title: Determination of the Duration of the Dual Antiplatelet Therapy by the Degree of the Coverage of The Struts on Optical Coherence Tomography From the Randomized Comparison Between Everolimus-eluting Stents Versus Biolimus A9-eluting Stents
Status: Not yet recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-1167
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Coronary Artery Disease
Keywords: Dual antiplatelet therapy duration; Optical coherence tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OCT-guided group: OCT-guided PCI with EES or BES
- Angiography-guidance group: Angio-guided PCI with EES or BES

SUMMARY:
This study is a retrospective and prospective follow-up study of patients who were participating in a randomized comparative study (DETECT-OCT trial) to determine the duration of dual antiplatelet therapy for neointimal hyperplasia after Biolimus stent and Everolimus stent insertion . The primary objective of this study was to determine the duration of double antiplatelet therapy (DAPT) based on OCT results at 3 months after percutaneous coronary intervention with OCT guide and percutaneous coronary intervention with guided angiography. After that, patients who were enrolled in the previous DETECT-OCT study will be followed up for a 10 years follow-up.

DETAILED DESCRIPTION:
This clinical trial will be followed for a long time until the 5th and 10th years of patients who have been registered for the DETECT-OCT study To assess the patient's status at 5- and 10-year, follow-up visits are scheduled at the outpatient visit if they are currently followed-up at the registry. However, if there is no follow-up observation at the current registrar, we will follow-up the telephone survey and visit as much as possible. Patients who have already passed the 5-year follow-up period from January 2, 2013, the first time to register, will be followed up by medical records to confirm the progress. To track the progress to the 10-year follow-up, we will conduct prospective observations by telephone survey.

ELIGIBILITY:
Inclusion Criteria:

* 1. patients who were enrolled in the previous DETECT-OCT study
* 2. Patients who agreed with informed consents

Exclusion Criteria:

* 1. Patients who disagreed with informed consents

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who already enrolled in DETECT-OCT
Sampling Method: Non-Probability Sample
Enrollment: 894 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival | At 5 years
  Free from death
Overall survival | At 10 years
  Free from death
Cardiac death | At 5 years
  Within 30 days after intervention, deaths due to myocardial infarction, cardiac perforation, tamponade or arrhythmia or death associated with intervention, death due to complications of intervention, and major cardiovascular deaths that can not be ruled out by a judgment of the screening adverse reaction review committee.
Cardiac death | At 10 years
  Within 30 days after intervention, deaths due to myocardial infarction, cardiac perforation, tamponade or arrhythmia or death associated with intervention, death due to complications of intervention, and major cardiovascular deaths that can not be ruled out by a judgment of the screening adverse reaction review committee.
Myocardial infarction | At 5 years
  (Non-Q-wave and Q-wave) due to occlusion of the target lesion or severe restenosis. The criteria for classification and diagnosis of myocardial infarction follow the Academic Research Consortium and the Third Universal Definition of MI. Coronary intervention Clinically significant myocardial infarction following the procedure has recently been defined by the Society for Cardiovascular Angiography and Interventions (SCAI)
Myocardial infarction | At 10 years
  (Non-Q-wave and Q-wave) due to occlusion of the target lesion or severe restenosis. The criteria for classification and diagnosis of myocardial infarction follow the Academic Research Consortium and the Third Universal Definition of MI. Coronary intervention Clinically significant myocardial infarction following the procedure has recently been defined by the Society for Cardiovascular Angiography and Interventions (SCAI)
Target lesion revascularization | At 5 years
  Repeatedly performing percutaneous intervention or target bypass repeatedly to the target lesion due to restenosis or other complications of the target lesion. The target lesion is defined as a treated segment of the vessel, ranging from 5 mm in the proximal portion of the stent to 5 mm in the distal portion of the stent.
Target lesion revascularization | At 10 years
  Repeatedly performing percutaneous intervention or target bypass repeatedly to the target lesion due to restenosis or other complications of the target lesion. The target lesion is defined as a treated segment of the vessel, ranging from 5 mm in the proximal portion of the stent to 5 mm in the distal portion of the stent.
Target vessel revascularization | At 5 years
  Repeatedly performing percutaneous intervention or target bypass repeatedly to the target vessel due to restenosis or other complications of the target vessel.
Target vessel revascularization | At 10 years
  Repeatedly performing percutaneous intervention or target bypass repeatedly to the target vessel due to restenosis or other complications of the target vessel.
Stent thrombosis | At 5 years
  Based on the Academic Research Consortium (ARC) definition.
  1. Definitive stent thrombosis
  2. Probable stent thrombosis
  3. Possible stent thrombosis
Stent thrombosis | At 10 years
  Based on the Academic Research Consortium (ARC) definition.
  1. Definitive stent thrombosis
  2. Probable stent thrombosis
  3. Possible stent thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Lee SY, Ahn CM, Yoon HJ, Hur SH, Kim JS, Kim BK, Ko YG, Choi D, Jang Y, Hong MK. Early Follow-Up Optical Coherence Tomographic Findings of Significant Drug-Eluting Stent Malapposition. Circ Cardiovasc Interv. 2018 Dec;11(12):e007192. doi: 10.1161/CIRCINTERVENTIONS.118.007192. PMID 30562088